CLINICAL TRIAL: NCT00339781
Title: Predictive and Protective Factors in the Cause of Diabetes: A Study in Twins
Brief Title: Predictive and Protective Factors in the Cause of Diabetes - A Study in Twins
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905109; 05-E-N109
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes; Type 1 Diabetes
Keywords: Fetomaternal Microchimerism; Cell Trafficking; Discordant Twins; Maternofetal Microchimerism; Diabetes Type I; Twins
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

SUMMARY:
This study, conducted at St. Bartholomew's Hospital, London, England, will determine whether cells passed from mother to offspring during pregnancy increase or decrease the child's risk of developing type 1 diabetes. Previous research has shown that certain cells that can be passed from mothers to their children during pregnancy may affect the child's chance of developing other autoimmune diseases. The cells from the mother may persist in the child's blood for years after birth and stimulate the child's immune system in such a way that may either increase or decrease the chance of the child developing diabetes. This study will determine whether these cells are present in identical twins, where only one of the twins has type 1 diabetes.

Participants in the British Diabetic Twins Study in England may be eligible to participate. Of each twin pair in the study, one must have type 1 diabetes and the other must be free of the disease. The twins' mother must be alive and willing to provide a blood sample. For female twins only, their children must be alive and willing to provide either a blood or a buccal cell sample (cheek swab).

Participants undergo the following procedures:

* Both twins in each twin pair provide a blood sample collected on a single occasion.
* The mother of each twin pair provides a blood sample collected on a single occasion.
* Children of female twins provide a single sample from either the mouth or blood. For children younger than 12 years of age, a cell sample is collected from the inside of the mouth (buccal) using a toothbrush. The child strokes the inside (cheek) of the mouth with the toothbrush ten times on each side, spits this into a collection vial, immediately rinses the mouth with water and adds this rinse to the sample collection vial. Children over 12 years of age may provide either a buccal cell sample or a blood sample.

DETAILED DESCRIPTION:
Type 1 diabetes is one of several autoimmune diseases of unclear etiology in which the discordance rate between identical twins is between 30-40%, even after many years of follow-up. This intermediate discordance rate indicates that there are clearly genetic factors at play in susceptibility to type 1 diabetes, with most genetic contribution coming from the HLA locus. However, this discordance rate also means that other, non-genetic factors, possibly environmental, lead to the development of disease in only one of two genetically identical individuals. No consensus exists on the nature of these putative environmental differences, which are all the more remarkable for occurring in twins that generally share the same intrauterine, family and school environment.

Recent evidence has suggested that the development of certain autoimmune diseases, particularly scleroderma, may be influenced by microchimerism: Both fetomaternal microchimerisms (persistence of fetal cells in the maternal circulation after birth of the child) and maternofetal microchimerism (persistence of maternal cells in the child's circulation for years after birth) have been suggested as creating an abnormal environment that might stimulate the development of autoimmunity in genetically susceptible individuals. The reverse is also possible, i.e., that these abnormal cells may stimulate the immune system in such a way that autoimmunity does not develop.

Identical or monozygotic (MZ) twins who are discordant for type 1 diabetes offer a unique experimental model in which to test the hypothesis that quantitative differences in persistent maternofetal microchimerism influence the development of type 1 diabetes in these genetically susceptible individuals. This study will use pairs of MZ twins discordant for the type 1 diabetes that are already participating in the British Diabetic Twins Study being conducted by Dr. David Leslie at St. Bartholomew's Hospital in London, UK. If the mothers of the twins (both female and male) and offspring of the female twins (only) are available for study, they will be asked to provide a single blood sample (twins, mothers, offspring greater than 12 years of age) or buccal cell sample (offspring less than or equal to 12 years of age) from which DNA will be purified. This is to confirm the origin of the chimeric cells; since cells are passed from the mothers to the offspring during pregnancy, we require (DNA) samples from the mothers of all twins (male and female) who participate in this study. But since the opposite is true, that cells can also be passed from offspring to their mothers during pregnancy, we will require (DNA) samples from the female twins' offspring to determine the true origin of any chimeric cells. The DNA will be used for HLA genotyping to identify nonshared HLA alleles that can be used to develop specific assays for the persistence of maternal DNA in the twins' circulation and quantitative PCR of the mother's genotype in CD3+ cells isolated from the twins. Since trafficking of chimeric cells can be bi-directional, twins who have had offspring of their own may have chimeric cells of both fetal and maternal origin in their circulation. To confirm the origin of the chimeric cells, the blood or buccal cells collected from the offspring of the twins will be genotyped and these compared to the genotypes of the twins' mothers. Blood will be drawn and DNA purified by Dr. Leslie's group in London; the genotyping and quantitative PCR will be performed by Dr. Artlett's group at Thomas Jefferson University, Philadelphia, which has been studying microchimerism since 1998. Results of the study may provide evidence in support of microchimerism as an influential factor in the development of type 1 diabetes. Evidence in support to this concept would be an important addition to the literature on "environmental" factors that influence type 1 diabetes etiology, and also suggest potential immunosuppression or other strategies in type 1 diabetes prevention.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA:

The twin subjects who are the focus of this study will be greater than or equal to 12 years of age and diabetes discordance must have been present for greater than 5 years.

The subjects must be able to understand and sign the informed consent documents, and thus severe mental incapacity is an exclusion criterion.

Female twins must not be currently pregnant or have had a miscarriage or abortion. Identical twin pairs (female or male) must not have undergone an organ or bone marrow transplantation, or a blood transfusion at any time in their lives.

There are no other health status criteria for participating in this study, except as noted above.

Patients may have other preexisting conditions.

There are no age limits for the offspring of the twins.

Subjects will not be excluded based on gender, ethnicity, race or religion.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240
Dates: Start 2005-02; Primary Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Bartholomew's Hospital, London, United Kingdom

REFERENCES:
- [Background] Tisch R, McDevitt H. Insulin-dependent diabetes mellitus. Cell. 1996 May 3;85(3):291-7. doi: 10.1016/s0092-8674(00)81106-x. No abstract available. PMID 8616883
- [Background] Christau B, Kromann H, Christy M, Andersen OO, Nerup J. Incidence of insulin-dependent diabetes mellitus (0--29 years at onset) in Denmark. Acta Med Scand Suppl. 1979;624:54-60. doi: 10.1111/j.0954-6820.1979.tb00719.x. PMID 284714
- [Background] Gottlieb MS, Root HF. Diabetes mellitus in twins. Diabetes. 1968 Nov;17(11):693-704. doi: 10.2337/diab.17.11.693. No abstract available. PMID 5687346